CLINICAL TRIAL: NCT01049893
Title: A Phase 1 Open-Label, Dose Finding, Safety and Tolerability Study of AC220 Administered Daily to Patients With Advanced Solid Tumors
Brief Title: Dose Finding, Safety and Tolerability Study for AC220 to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC220-004
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — quizartinib; Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC220 (Experimental): Dose finding study. Number of arms dependant upon dose limiting toxicities.
  Interventions: Drug: Compound AC220

INTERVENTIONS:
Drug: Compound AC220 — Precomplexed powder in bottle formulation supplied as 135 mg in a 60 cc polyethylene terephthalate (PET) plastic bottle. Requires reconstitution by a pharmacist, must be stored securely, and protected from light.
  Other Names: AC010220 * 2HCl, oral powder for reconstitution

SUMMARY:
AC220 will be administered as a once daily oral solution given continuously as 28-day treatment cycles, without food and without any rest periods, as long as there is no evidence of disease progression or unacceptably severe adverse events (AEs) related to the study drug.

DETAILED DESCRIPTION:
A phase 1 open-label, dose finding study of AC220 in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age ≥18 years
2. Understand and voluntarily sign the informed consent form for this study
3. Available for periodic follow-up at the investigative site
4. Able to swallow the liquid study drug
5. ECOG performance status of 0 - 2
6. Histological diagnosis of a primary solid tumor malignancy that meets the following criteria:

   * Evidence (radiographic or tissue confirmation) that the disease is metastatic (locally advanced disease is allowable only if no surgical or local therapeutic option exists); and
   * Disease which has progressed on or following currently available standard therapies or for which no curative therapy exists (Prior adjuvant, neoadjuvant, and investigational therapies are permitted.)
7. Measurable disease by computer tomography (CT) or magnetic resonance imaging (MRI) scans per RECIST.
8. Prior anticancer therapy, radiotherapy, hormonal, and immunotherapy are allowed. Patients must have recovered from toxicity of prior therapy (ie, toxicity has resolved to Grade 1, or to pre-treatment baseline, or is deemed irreversible). At least 4 weeks must have elapsed since the last systemic therapy (6 weeks for nitrosoureas, mitomycin-C, and liposomal doxorubicin), immunotherapy, or radiotherapy and the beginning of study drug administration. For participants with GIST on approved tyrosine kinase inhibitors (TKI), at least 2 weeks must have elapsed since the last dose of TKI.
9. Adequate bone marrow function, defined as:

   * Absolute neutrophil count (ANC) (neutrophils and bands) ≥1.5 x 10^9 cells/L
   * Platelet count ≥ 100 x 10^9 cells/L
   * Hemoglobin ≥ 9.0 g/dL
10. Adequate hepatic function, defined as:

    * Total serum bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x the institutional ULN
11. Adequate renal function, defined as:

    * Serum creatinine ≤ 1.5 x the institutional ULN
12. Prothrombin time or partial thromboplastin time (PT- PTT) ≤ 1.5 x the ULN
13. Serum potassium, magnesium, and calcium levels should be at least within institutional normal limits, and every effort should be made to keep potassium concentrations above 4.0 mEq/dL, magnesium concentrations above 1.8 mg/dL, and serum calcium at normal concentration with the administration of oral/IV potassium and/or magnesium and/or calcium replacement during the study. If this is not possible, potassium and magnesium (and calcium) concentrations should at least be kept within institutional normal limits.
14. Fully recovered (≤ Grade 1 or returned to baseline or deemed irreversible) from the acute effects of prior cancer therapy before initiation of study drug administration.
15. Baseline left ventricular ejection fraction (LVEF) ≥ 45% (or ≥ institutional lower limit of normal if institutional lower limit of normal is below 45%) as assessed by 2-dimensional ECHO or MUGA as per institutional practice. If repeat LVEF assessment is required, the same modality should be used throughout the duration of study, whenever possible.
16. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 3 months after the study in such a manner that the risk of pregnancy is minimized. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not post menopausal (defined as amenorrhea > 12 consecutive months; or who is on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL). Additionally, premenopausal women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, are practicing abstinence, or whose partner is sterile (eg, vasectomy), should be considered to be of childbearing potential.
17. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 72 hours prior to the start of study drug.

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable contraceptive method to avoid pregnancy for the entire study period and for at least 3 months after the study.
2. Women who are pregnant or breastfeeding
3. WOCBP with a positive pregnancy test on enrollment prior to study drug administration
4. Men who are unwilling or unable to use an acceptable method of birth control if their sexual partners are WOCBP for the entire study period and for at least 3 months after completion of the study
5. Patients with known untreated, symptomatic or uncontrolled brain or central nervous system (CNS) metastases. Patients with treated brain or CNS metastases that are radiographically stable for 3 months or longer are eligible.
6. A serious uncontrolled medical disorder or active infection which would impair the ability of the patient to receive study drug
7. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within 12 months prior to study entry
   * Uncontrolled angina within 6 months prior to study entry
   * Congestive heart failure (CHF) New York Heart Association (NYHA) class 3 or 4, or patients with history CHF NYHA class 3 or 4 in the past, unless the screening ECHO or MUGA within 14 days prior to study entry results in a LVEF that is ≥ 45% (or ≥institutional lower limit of normal)
   * Diagnosed or suspected congenital long QT syndrome
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes [TdP])
   * Prolonged QTc interval on pre-entry ECG (≥ 450 ms)
   * Any history of second or third degree heart block
   * Uncontrolled hypertension
   * Obligate need for a cardiac pacemaker
   * Complete left bundle branch block
   * Atrial fibrillation
8. Known infection with human immunodeficiency virus (HIV)
9. Known active hepatitis A, B, or C or other active liver disease
10. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent
11. Investigational agents during or within 4 weeks prior to the start of study drug
12. Use of drugs that are generally accepted to have a risk of causing prolonged QTc and/or TdP and/or are CYP3A4 inhibitors. Patients who have discontinued any of these medications must have a washout period of at least 5 days or at least 5 half-lives of the drug (whichever is greater) prior to the first dose of study drug and should not be allowed to take these medications during the study drug dosing.
13. Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the judgment of the Principal Investigator or Sponsor, could jeopardize patient safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AC220 given once daily without food continuously for 28 days (1 cycle) to patients with advanced solid tumors. | Repeatedly measured at multiple timepoints during 1st cycle; every 2 weeks thereafter

SECONDARY OUTCOMES:
Pharmacokinetic (PK) and pharmacodynamic (PD) parameters of AC220 in this patient population under the conditions of the study, including a careful and detailed evaluation of the ECG effects of AC220 in relation to plasma drug concentration | Repeatedly measured at multiple timepoints during the first cycle of treament.
Preliminary evidence of antitumor biology or clinical activity of AC220 in patients enriched for diseases whose pathophysiology is directly related to aberrant c-KIT receptor or platelet-derived growth factor receptor signaling. | Measured every 28 days (per treatment cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Gammon, MB BS, MRCP, Study Director — Interim Chief Medical Officer, Ambit Biosciences Corporation
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Papadopoulos KP, Ben-Ami E, Patnaik A, Trone D, Li J, Demetri GD. Safety and tolerability of quizartinib, a FLT3 inhibitor, in advanced solid tumors: a phase 1 dose-escalation trial. BMC Cancer. 2018 Aug 6;18(1):790. doi: 10.1186/s12885-018-4692-z. PMID 30081867